CLINICAL TRIAL: NCT01398553
Title: Armeo® Versus Standard Physiotherapy for Upper Limb Rehabilitation in Patients With Acquired Brain Lesions
Brief Title: Automated Versus Standard Physiotherapy for Upper Limb Rehabilitation in Patients With Acquired Brain Lesions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the human resources in the organisation are to limited to do the trial
Sponsor: Krankenhaus Bozen (Other)
Collaborators: Valduce Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gesundheitsbezirk Bozen
Record Dates: First submitted 2010-11-29; First posted 2011-07-20 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Vascular Accident, Brain; Traumatic Brain Injury
Keywords: stroke; tbi; rehabilitation; upper limb
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armeo Spring (Experimental)
  Interventions: Device: Armeo Spring
- conventional physiotherapy (Active Comparator)
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Device: Armeo Spring — 30min Armeo Spring + 15min task oriented therapy over 6 weeks Frequency: 3 x/week
  Other Names: group A
  Arms: Armeo Spring
Other: conventional physiotherapy — 30min occupational therapy(15min ADL-training, 15min repetitive training) + 15min task oriented therapy over 6 weeks Frequency: 3x/week
  Other Names: group B
  Arms: conventional physiotherapy

SUMMARY:
The Armeo Spring has proven its effectiveness in the rehabilitation of acute stroke patients. It neutralizes limb weight, enabling patients to use residual control in both arm and hand and to follow exercises guided by simulations of real-life challenges. The Armeo Spring incorporates wrist pronation and supination, allowing patients to enhance functional reaching patterns.

Aim of the study is to compare the Armeo device with standard physiotherapy in chronic patients with acquired brain lesions.

The result of the trial should show which treatment is more effective in the clinical practice. A significant better outcome of one arm should suggest to follow one treatment strategy more than the other.

ELIGIBILITY:
Inclusion Criteria:

* 6 month after the onset of disease
* acquired brain lesions in adults with upper limb hemiparesis
* modified Ashworth <= 3
* muscular strength MRC =>1 mano; MRC =>2 elbow e shoulder
* Fugl Meyer => 18

Exclusion Criteria:

* NYHA >III
* MMSE (mini mental status examination test) < 24
* muscular strength (MRC) < 1
* Dystonia, spasticity (Ashworth => 3)
* articular contractions in the upper limb
* previous upper limb lesions
* cognitive/language impairment likely to influence assessments
* any diagnosis likely to interfere with rehabilitation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Score for sensorymotor recovery of the upper limb after stroke | Enrollment
Fugl Meyer Score for sensorymotor recovery of the upper limb after stroke | Baseline
Fugl Meyer Score for sensorymotor recovery of the upper limb after stroke | 6 weeks
Fugl Meyer Score for sensorymotor recovery of the upper limb after stroke | 8 weeks
Fugl Meyer Score for sensorymotor recovery of the upper limb after stroke | 12 weeks

SECONDARY OUTCOMES:
Upper Extremity Motor Activity Log for measuring real use of the upper limb | Enrolment
Upper Extremity Motor Activity Log for measuring real use of the upper limb | Baseline
Upper Extremity Motor Activity Log for measuring real use of the upper limb | 6 weeks
Upper Extremity Motor Activity Log for measuring real use of the upper limb | 8 weeks
Upper Extremity Motor Activity Log for measuring real use of the upper limb | 12 weeks
Wolf Motor Function Test for measurement of timed joint-segment movements | Enrolment
Wolf Motor Function Test for measurement of timed joint-segment movements | Baseline
Wolf Motor Function Test for measurement of timed joint-segment movements | 6 weeks
Wolf Motor Function Test for measurement of timed joint-segment movements | 8 weeks
Wolf Motor Function Test for measurement of timed joint-segment movements | 12 weeks
Clinical Global Impression Score for the measurement of change over time of the illness' severity | Enrolment
Clinical Global Impression Score for the measurement of change over time of the illness' severity | Baseline
Clinical Global Impression Score for the measurement of change over time of the illness' severity | 6 weeks
Clinical Global Impression Score for the measurement of change over time of the illness' severity | 8 weeks
Clinical Global Impression Score for the measurement of change over time of the illness' severity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zelger, MD, Principal Investigator — Krankenhaus Bozen; Franco Molteni, MD, Study Director — Valduce Hospital; Elisabeth Hofer, MD, Study Chair — Krankenhaus Bozen; Mauro Rossini, MSc, Study Chair — Valduce Hospital
Locations (2):
- Italy (2):
  - Valduce Hospital, Costa Masnaga, Lombardy
  - Krankenhaus Bozen, Bolzano, Südtirol

REFERENCES:
- [Background] Kwakkel G, Kollen BJ, Krebs HI. Effects of robot-assisted therapy on upper limb recovery after stroke: a systematic review. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):111-21. doi: 10.1177/1545968307305457. Epub 2007 Sep 17. PMID 17876068
- [Background] Prange GB, Jannink MJ, Groothuis-Oudshoorn CG, Hermens HJ, Ijzerman MJ. Systematic review of the effect of robot-aided therapy on recovery of the hemiparetic arm after stroke. J Rehabil Res Dev. 2006 Mar-Apr;43(2):171-84. doi: 10.1682/jrrd.2005.04.0076. PMID 16847784
- [Background] Lam P, Hebert D, Boger J, Lacheray H, Gardner D, Apkarian J, Mihailidis A. A haptic-robotic platform for upper-limb reaching stroke therapy: preliminary design and evaluation results. J Neuroeng Rehabil. 2008 May 22;5:15. doi: 10.1186/1743-0003-5-15. PMID 18498641
- [Background] Masiero S, Celia A, Rosati G, Armani M. Robotic-assisted rehabilitation of the upper limb after acute stroke. Arch Phys Med Rehabil. 2007 Feb;88(2):142-9. doi: 10.1016/j.apmr.2006.10.032. PMID 17270510
- See also: Participating Centre — http://www.valduce.it